CLINICAL TRIAL: NCT02633007
Title: A Phase 1 Study of the Safety and Pharmacokinetics (PK) of Levodopa Following Administration of CVT 301 (Levodopa Inhalation Powder) in Adults With Asthma
Brief Title: A Study of the Safety and Pharmacokinetics of Levodopa Following Administration of CVT 301 (Levodopa Inhalation Powder) in Adults With Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CVT-301-008
Record Dates: First submitted 2015-12-11; First posted 2015-12-17 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Carbidopa

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- CVT-301 then Placebo (AB) (Experimental): All subjects will receive both CVT-301 and placebo in two dosing periods separated by one day. Subjects will be randomized 1:1 into sequence AB or BA [CVT-301 (A) administered first, followed by placebo (B), or the reverse order (BA)] and they will start pre-treatment of carbidopa (as Lodosyn®) administered every 8 hours until the completion of all study treatments.
  Interventions: Drug: CVT-301 (levodopa inhalation powder); Drug: Carbidopa; Other: Placebo
- Placebo then CVT-301 (BA) (Experimental): All subjects will receive both CVT-301 and placebo in two dosing periods separated by one day. Subjects will be randomized 1:1 into sequence AB or BA [CVT-301 (A) administered first, followed by placebo (B), or the reverse order (BA)] and they will start pre-treatment of carbidopa (as Lodosyn®) administered every 8 hours until the completion of all study treatments.
  Interventions: Drug: CVT-301 (levodopa inhalation powder); Drug: Carbidopa; Other: Placebo

INTERVENTIONS:
Drug: CVT-301 (levodopa inhalation powder) — Capsules containing l-dopa, designed to deliver ldopa to the lung using the CVT-301 inhaler. CVT-301 will be administered 3 times, 4 hours apart, and 1 hour following the administration of carbidopa.
Drug: Carbidopa — Administered orally according to the carbidopa dosing schedule.
  Other Names: Lodosyn ®
Other: Placebo — Placebo of CVT-301 is administered in the same way as the investigational product, except that it does not contain l-dopa.

SUMMARY:
This study is a double-blind, randomized, placebo-controlled, 2-period, crossover study to evaluate safety and PK of 3 doses of CVT 301 levodopa (l-dopa) in adults with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects will be men or women in good general health with a diagnosis of mild or moderate asthma;
* On a stable regimen of asthma medications for at least 30 days prior to screening;
* Body mass index (BMI) 18 to 32 kg/m2;
* Forced expiratory volume in one second (FEV1) ≥60% of predicted for race, age, sex, and height;
* FEV1/FVC (forced vital capacity) ratio ≥70%.

Exclusion Criteria:

* More than 2 hospitalizations or emergency room visits, or more than 3 courses of systemic steroids in the past 12 months or 1 course within the past 8 weeks for respiratory illness;
* Asthma exacerbation within 8 weeks before screening;
* Unscheduled or urgent visit to any medical facility for asthma-related problems within 8 weeks before screening;
* History of intubation or intensive care unit admission for asthma in the past 5 years;
* History of chronic obstructive pulmonary disorder (COPD) requiring intermittent or continuous use of any oral or inhaled medication therapy within last 3 years;
* Renal impairment as defined by a calculated creatinine clearance of ≤ 80 mL/minute.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-12; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in pulmonary function | within 90 min prior to dose administration and specified time points up to 24 hours after first inhalation
  Pulmonary function will be measured by spirometry using the guideline specified by the Third National Health and Nutrition Examination Survey (NHANES III)

SECONDARY OUTCOMES:
Number of subjects with Adverse Events (AEs) including Serious AEs | up to 12 days
Maximum observed plasma drug concentration (Cmax) | within 30 min prior to first CVT-301 dose administration and specified time points up to 24 hours post-dose
Time to maximum observed plasma drug concentration (Tmax) | within 30 min prior to first CVT-301 dose administration and specified time points up to 24 hours post-dose
Area under the concentration time curve over the dosing interval (AUC0-last) | within 30 min prior to first CVT-301 dose administration and specified time points up to 24 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Harald Murck, MD, PhD, Study Director — Acorda Therapeutics
Locations (3):
- United States (3):
  - Site 002, Daytona Beach, Florida
  - Site 001, North Dartmouth, Massachusetts
  - Site 003, Dallas, Texas